CLINICAL TRIAL: NCT02861092
Title: Antibiotic-related Serious Adverse Events in Obese Patients Treated for Bone and Joint Infection
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0537
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
Keywords: Serious adverse event; bone and joint infection; obesity; dose adjustment
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It exists recommendations to get an optimal antibiotic treatment for bone and joint infection and prescription of antibiotics in the bone and joint infections on material meets certain obligations: the micro-organism must be known, the antibiotic therapy must be started in association, obtaining high plasma levels, use of molecules having good bone circulation. It is recommended to initially administer treatment with intravenous route and to propose an oral relay, under conditions. It is recommended to administer the antibiotic treatment for at least 6 weeks.

The dosages of antibiotics are adapted to the weight of patients in order to respond to those recommendations. But little is known about the optimal dose of treatment to give to obese patients (BMI>=30) and the frequency of serious adverse events in these patients in which the dosage is then higher can be more important compared to non-obese patients. The aim of the study is then to evaluate the risk of occurrence of serious adverse events in obese patients and to identify risks factors.

This study consists in a retrospective cohort of obese patients treated for a bone or joint infection and having had a serious adverse event. Several data are collected concerning: demographics data, treatment responsible of the serious adverse event (molecules, dosage, route), description of the serious adverse event, residual rate for vancomycin.

ELIGIBILITY:
Inclusion Criteria:

* patients (i.e age ≥ 15 year-old) with bone and joint infection
* with or without implant
* for which the BMI is >=30
* having had a serious adverse event related to the antibiotic treatment.

Exclusion Criteria:

* none

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Obese patients, under antibiotic treatement for bone or joint infection and who presented a serious adverse event
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Description of all serious adverse events observed in obese patients and non-obese patients | The patients included have presented a serious adverse event between 2008 and 2015
  The data concerning the serious adverse events are collected in this Cohort. It is molecule, dosage, description of the adverse event. A severity grade is allocated to every adverse event, based on the " Common Terminology Criteria for Adverse Events ". This is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term (from 1 to 5). Serious adverse events have a grade >=3. This description will highlight particular the antibiotics the most implicated in serious adverse events

SECONDARY OUTCOMES:
Analysis of accountability of the antibiotics in serious adverse events in obese patients | The patients included have presented a serious adverse event between 2008 and 2015.
  A comparison of the serious adverse events is made between the group of obese patients, a group of non-obese patients treated for bone and joint infection and a group of obese patients treated for bone and joint infection but who had never had an adverse event. The role of the vancomycin in the serious adverse event will be compared in the 3 populations where the lean body mass (total mass of the skin, bones, muscles, organs and fluids of the human body), the fat body mass and the total mass will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, MD PhD, Principal Investigator — Centre de référence des infections ostéo-articulaires
Locations (1):
- Centre de référence des infections ostéo-articulaires, Hôpital de la Croix-Rousse, 103 Grande Rue de la Croix-Rousse,, Lyon, France

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr